CLINICAL TRIAL: NCT05443048
Title: Evaluation of Monolithic Milled Complete Removable Dentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frauke Müller (Other)
Responsible Party: Sponsor-Investigator, Frauke Müller, Professor, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ivotion Pilot Study
Record Dates: First submitted 2022-06-21; First posted 2022-07-05 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2022-06

CONDITIONS: Complete Edentulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivoclar Ivotion Denture System (Experimental)
  Interventions: Device: Ivoclar Ivotion Denture System

INTERVENTIONS:
Device: Ivoclar Ivotion Denture System — Fabrication of maxillary and mandibular complete removable dental prosthesis with the Ivoclar Ivotion Denture System

SUMMARY:
The use of complete removable dental prostheses (CRDP) is a reliable and effective treatment option for the rehabilitation of edentulous persons.

In recent years, the use of computer-aided design/computer-aided manufacturing (CAD/CAM) methods has become more popular for the fabrication of CRDPs, including subtractive methods (milling) from a prefabricated resin puck. They present various advantages compared to conventional fabrication methods, namely improved mechanical properties, superior surface characteristics, shortened manufacturing time and lower cost for the patient.

However, one of the shortcomings in the manufacturing of CRDPs from a single block of resin is obtaining an adequate esthetic outcome, as the transition between the gingiva-colored (pink) and tooth-colored (white) resin is not as precise as with prefabricated prosthetic teeth which are incorporated into a denture base. A novel technology has recently been launched on the market and includes a new design of distribution of pink and white resin inside a prefabricated resin puck, which would allow a superior esthetic outcome than previous techniques.

The aim of this pilot study is to assess the end result of one of the available systems used for fabricating digital dentures (Ivoclar® Digital Denture®), while using the corresponding monolithic resin puck (Ivoclar® Ivotion Denture System®), and therefore determining whether this new technique is an adequate option for treating edentulous patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed Consent as documented by signature
* Healed edentulous maxilla and mandible (minimum one year since last extraction)

Exclusion Criteria:

* Contraindications to the medical devices used, e.g. known hypersensitivity or allergy
* Vulnerable subjects
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the investigation
* Participation in another investigation with a MD in the field of dentistry
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Reported severe bruxism or clenching habits, clinically present oro-facial pain
* Width of edentulous maxilla > 80 mm
* Width of edentulous mandible > 80 mm
* Vertical height needed for maxillary prosthesis > 38 mm
* Vertical height needed for mandibular prosthesis > 38 mm
* Depression: Geriatric Depression Scale > 9
* Xerostomia: SSFR ≤ 0.7ml/min
* Dementia: Clock-Drawing Test ≤ 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Esthetics | Baseline (BL, with existing dentures)
  The transition between the pink and white resin will be evaluated by means of a Visual Analogue Scale esthetic score Maximum (best outcome): 1000 Minimum (worst outcome): 0
Esthetics | Day 0 (T0, new dentures)
  The transition between the pink and white resin will be evaluated by means of a Visual Analogue Scale esthetic score Maximum (best outcome): 1000 Minimum (worst outcome): 0
Esthetics | 3 months (T1)
  The transition between the pink and white resin will be evaluated by means of a Visual Analogue Scale esthetic score Maximum (best outcome): 1000 Minimum (worst outcome): 0

SECONDARY OUTCOMES:
Oral health-related quality of life | Baseline (BL, with existing dentures)
  OHIP-EDENT: validated questionnaire with 19 questions related to 7 dimensions, by means of a 6-item Likert scale Maximum (worst outcome): 7 Minimum (best outcome: 0
Oral health-related quality of life | Day 0 (T0, new dentures)
  OHIP-EDENT: validated questionnaire with 19 questions related to 7 dimensions, by means of a 6-item Likert scale Maximum (worst outcome): 7 Minimum (best outcome: 0
Oral health-related quality of life | 3 months (T1)
  OHIP-EDENT: validated questionnaire with 19 questions related to 7 dimensions, by means of a 6-item Likert scale Maximum (worst outcome): 7 Minimum (best outcome: 0
Denture satisfaction | Baseline (BL, with existing dentures)
  Denture Satisfaction Index: validated questionnaire with 24 questions related to 9 dimensions, by means of a Visual Analogue Scale Maximum (best outcome): 900 Minimum (worst outcome): 0
Denture satisfaction | Day 0 (T0, new dentures)
  Denture Satisfaction Index: validated questionnaire with 24 questions related to 9 dimensions, by means of a Visual Analogue Scale Maximum (best outcome): 900 Minimum (worst outcome): 0
Denture satisfaction | 3 months (T1)
  Denture Satisfaction Index: validated questionnaire with 24 questions related to 9 dimensions, by means of a Visual Analogue Scale Maximum (best outcome): 900 Minimum (worst outcome): 0
Masticatory analysis | Baseline (BL, with existing dentures)
  Chewing efficiency will be evaluated with a two-color mixing ability test
Masticatory analysis | Day 0 (T0, new dentures)
  Chewing efficiency will be evaluated with a two-color mixing ability test
Masticatory analysis | 3 months (T1)
  Chewing efficiency will be evaluated with a two-color mixing ability test
Prosthetic Evaluation | Day 0 (T0, new dentures)
  Denture quality objectively based on the seven criteria adopted from Alfadda et al., 2014, using a scoring sheet with 16 questions, by means of a 3-item Likert scale Maximum (worst score): 48 Minimum (best score): 16
Prosthetic Evaluation | 3 months (T1)
  Denture quality objectively based on the seven criteria adopted from Alfadda et al., 2014, using a scoring sheet with 16 questions, by means of a 3-item Likert scale Maximum (worst score): 48 Minimum (best score): 16
Number of prosthetic maintenance needed | 3 months (T1)
  events such as adjustment and repair requirements will be recorded
Willingness to Pay | 3 months (T1)
  open-ended contingency valuation (CV) method of questioning with the use of a payment card. The score is the amount in Swiss Francs the participant would be willing to pay for the treatment.
  Maximum: no maximum Minimum: 0.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Maniewicz, Dr, Principal Investigator — Research and Teaching Fellow
Locations (1):
- University of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No